CLINICAL TRIAL: NCT04891289
Title: A Randomized Phase II Study of Systemic Chemotherapy With or Without HAI FUDR/Dexamethasone in Patients With Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Gemcitabine and Oxaliplatin Chemotherapy With or Without a Floxuridine and Dexamethasone Pump in People With Cholangiocarcinoma That Cannot Be Removed With Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-348
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Gemcitabine; Oxaliplatin; Floxuridine; Dexamethasone Pump; 20-348
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Oxaliplatin; Dexamethasone; Floxuridine

STUDY DESIGN:
Intervention Model Description: This is a multi-center, prospective randomized controlled phase II study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- HAI FUDR plus GemOx (Arm 1) (Experimental): Surgical HAI pump placement. 2. HAI FUDR [(0.12 mg/kg/day) x wt (kg) x (30ml) / pump flow rate ] and dexamethasone [1 mg/day * 30] / pump flow rate ] on Day 1 of each cycle. Chemotherapy with HAI FUDR/Dex will commence no sooner than 14 days postsurgical placement of HAI pump. 3. Gemcitabine (800 mg/m2 IV over 30 minutes) and oxaliplatin (85 mg/ m2 IV over 120 minutes on Days 1 and 15 of each cycle; however, for patients in Arm 1, initiation of systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement, so the first dose of systemic chemotherapy will be given on Cycle 1, Day 15, and then every 2 weeks thereafter.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Dexamethasone; Drug: Floxuridine (FUDR); Device: Implanted Medical Device
- GemOx alone (Arm 2) (Active Comparator): Gemcitabine (800 mg/m2 IV over 30 minutes) and oxaliplatin (85 mg/m2 IV over approximately 120 minutes) on Days 1 and 15 of each 28-day cycle.For patients in Arm 2, systemic therapy will be administered on Days 1 and Day 15 of each Cycle on a 28-day cycle basis, compromised of Gemcitabine and Oxaliplatin. If a patient randomized to Arm 2 has intrahepatic progression on any follow-up scan during study treatment, that patient will be eligible to crossover to Arm 1 and commence to pump placement surgery and HAI FUDR treatment. Patients with any extrahepatic progression will not be eligible to utilize the crossover arm. Arm 2 patients will have 28 days from date of the scan showing intrahepatic progression to proceed to the crossover arm.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — See arm for details.
Drug: Oxaliplatin — See arm for details.
Drug: Dexamethasone — See arm for details.
  Arms: HAI FUDR plus GemOx (Arm 1)
Drug: Floxuridine (FUDR) — See arm for details.
  Arms: HAI FUDR plus GemOx (Arm 1)
Device: Implanted Medical Device — Implanted hepatic arterial infusion pump by surgical oncology, to deliver HAI therapy
  Arms: HAI FUDR plus GemOx (Arm 1)

SUMMARY:
This study will compare the safety and effects of HAI floxuridine and dexamethasone combined with the standard chemotherapy drugs gemcitabine and oxaliplatin (GemOx) with those of GemOx alone in people with untreated cholangiocarcinoma that cannot be removed with surgery. The researchers want to find out whether the study treatment works better than the standard chemotherapy to delay progression of disease. For the study treatment to be considered better than the standard treatment, the study treatment should increase the time until progression of disease by an average of 3 months, compared with the usual approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ECOG 0-1
* Histologically confirmed intrahepatic cholangiocarcinoma (also variously reported as peripheral cholangiocarcinoma, cholangiolar carcinoma or cholangiocellular carcinoma) (IHC). Confirmation of the diagnosis at MSKCC or at the enrolling institution must be obtained prior to randomization.
* Clinical or radiographic evidence of metastatic disease confined to the liver. Note: presence of regional (porta hepatis) lymph node metastases will be allowed, provided they are amenable to resection. (Note: If peritoneal or other extrahepatic disease is found at time of pump placement, the pump will not be implanted. The patient will be removed from study, deemed nonevaluable and will not count toward the overall study accrual.)
* Radiographically measurable disease. Measurable disease is defined as disease that can be assessed with 2-dimensional measurements on a cross-sectional imaging. Minimum lesion size is 2 cm in greatest diameter as per RECIST criteria.
* Disease must be considered unresectable at the time of preoperative evaluation.*
* Considered candidate for general anesthesia, abdominal exploration and hepatic artery pump placement.
* Patients with chronic hepatitis and/or cirrhosis are eligible, but must be Child-Pugh class A.
* WBC ≥ 2,000/mcL , ANC ≥ 1000/mcL
* Platelet count ≥ 75,000/mcL
* Creatinine ≤ 1.8 mg/dL
* Total bilirubin < 1.5 mg/dL
* Hgb > 7 g/dL The % involvement of the liver will be determined by radiologists after review of imaging

Exclusion Criteria:

* Presence of distant metastatic disease. Patients will undergo radiographic evaluation to exclude the possibility of distant metastatic disease. For patients who have undergone pre- or post-operative biopsies that definitively diagnose IHC, the diagnostic studies may be modified at the discretion of the MSKCC Principal Investigator. Clinical or radiographic evidence of metastatic disease to regional lymph nodes will be allowed, provided it is amenable to resection.
* Patients previously treated with systemic chemotherapy for IHC will be non-eligible.
* Prior treatment with FUDR.
* Prior external beam radiation therapy to the liver.
* Prior ablative therapy to the liver.
* Diagnosis of sclerosing cholangitis.
* Clinical evidence or portal hypertension (ascites, gastroesophageal varices, or portal vein thrombosis; surgically related ascites does not exclude the patient).
* Active infection within one week prior to HAI placement.
* Pregnant or lactating women.
* History of other malignancy within the past 3 years except with early stage/localized cancer that was surgically resected or radiation treatment that would yield the same result as surgery within the past 3 years.
* Life expectancy <12 weeks.
* Inability to comply with study and/or follow-up procedures.
* History of peripheral neuropathy. There is no exclusion of patients based on sex, ethnicity or race. For these reasons, the study results are expected to be generalizable to the Medicare beneficiary population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
assess progression-free survival (PFS) | 2 years
  will be done using RECIST (version 1.1).

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (10):
  - National Heart, Lung, and Blood Institute (NIH) (Data Collection Only), Bethesda, Maryland
  - Washington University (Data Collection Only), St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge - Limited Protocol Activities, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth - Limited Protocol Activities, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen - Limited Protocol Activities, Montvale, New Jersey
  - Memorial Sloan Kettering Commack - Limited Protocol Activities, Commack, New York
  - Memorial Sloan Kettering Westchester - Limited Protocol Activities, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau - Limited Protocol Activities, Uniondale, New York
  - Duke University (Data Collection Only), Durham, North Carolina
- Erasmus University (Data Collection Only), Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm